CLINICAL TRIAL: NCT03874130
Title: Open-label, Dose-escalating, Non-randomized, Single-Center Study to Determine the Safety and Pharmacokinetic Profiles of Scopolamine in Healthy Volunteers
Brief Title: Scopolamine in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Repurposed Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DPI-386-DE-10
Record Dates: First submitted 2018-12-13; First posted 2019-03-14 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2019-12

CONDITIONS: Major Depressive Disorder (MDD)
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Scopolamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Scopolamine (Active Comparator): 0.2 mg scopolamine HBr per dose
  Interventions: Drug: Scopolamine
- IV Scopolamine (Active Comparator): 4.0 μg/kg; 15 minute IV infusion
  Interventions: Drug: Scopolamine

INTERVENTIONS:
Drug: Scopolamine — IV Scopolamine
  Other Names: scopolamine HBr

SUMMARY:
This single-site clinical trial is an open-label study to identify the safety and pharmacokinetics of DPI-386 Nasal Gel (intranasal scopolamine gel) and IV Scopolamine. The study will require subjects to receive either multiple doses of 0.2 mg or a single dose of 0.4 mg, 0.6 mg, 0.8 mg, 1.0 mg, or 1.2 mg of DPI-386 Nasal Gel or 0.4 mg/mL IV Scopolamine per the assigned treatment cohort. Multiple PK blood draws will be collected dependent on cohort assignment. Vital signs and ECGs will be collected. No efficacy will be tested. Subjects will be monitored for at least eight hours after the final dose. There could be up to 160 subjects enrolled stratified equally by gender.

Screening will not occur until after subjects have signed the informed consent form (ICF). Screening will include hematology, biochemistry, urinalysis, alcohol and drug screen, physical examination, including vital signs and ECG, and review of medical history by the PI or qualified designee, serum pregnancy test as applicable, and agreement to adhere to the study lifestyle requirements.

Subject data will be recorded in the source documents and appropriate eCRF.

DETAILED DESCRIPTION:
The investigational product is a combination product comprised of: (a) a vial prefilled with DPI-386 Nasal Gel, and (b) a nasal gel pump attached to the vial during the manufacturing process. For Cohorts 1 through 4, 9 through 10,13, and 14 each 0.12 gram of the gel contains 0.2 mg of scopolamine HBr as the active ingredient along with the excipients sodium citrate, citric acid, sodium metabisulfite, glycerin, benzalkonium chloride, polyvinyl alcohol and purified water. For Cohorts 1 through 4, 9, 10 and 13 through 16 each vial of DPI-386 Nasal Gel is a multi-dose product, sufficient for six individual doses. Each pumping action is designed to deliver a single 0.12 g dose. The DPI-386 Nasal Gel for Cohorts 1 through 4, 13 and 14 is formulated to contain 0.2 mg scopolamine HBr per 0.12 g dose, with each dose therefore described as "0.2 mg / 0.12 g". For Cohort 6 the dose is "0.8 mg / 0.12 g", and for cohort 7 the dose is "1.0 mg / 0.12 g", and for Cohort 8 the dose is "1.2 mg / 0.12 g", and for Cohort 11 the dose is "0.4 mg / 0.12 g", and for Cohort 12 and 15 the dose is "0.6 mg / 0.12 g", delivered in a single dose, and for Cohort 16 the dose is "0.6 mg / 0.12 g", in a modified excipient formulation, delivered in a single dose.

For Cohort 16 only: Each 0.12 gram of the gel contains 0.6 mg of scopolamine HBr as the active ingredient along with a modified formulation of excipients sodium citrate, citric acid, sodium metabisulfite, glycerin, benzalkonium chloride 100, polyvinyl alcohol 18, and purified water.

Each vial/pump unit must be primed by research staff prior to first dose delivery. Subjects will self-administer the drug under guidance from the study staff.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated ICF.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Male or female, aged 18 to 40 (inclusive).
4. Males and females must agree to use highly effective contraception (e.g. double barrier method) for 4 weeks after receiving the last dose of treatment.
5. Have a body mass index (BMI) within a range of 18 to 30 inclusive.
6. In good general health as evidenced by medical history with no recent history or current diagnosis of significant cardiovascular or respiratory problems as assessed by the PI or qualified designee.
7. Hematology, biochemistry, urinalysis and drug and alcohol laboratory test results that are determined by the PI or qualified designee to be not clinically significant.
8. Ability to take intranasal medication (for Cohorts 1-4, and 6-15 only) and willingness to adhere to the study schedule and time constraints.
9. For females of child-bearing potential: willingness to provide a sample for the pregnancy test upon every visit. Test must be negative.

   Note: Women of non-childbearing potential are defined as those who are non-surgically sterile (i.e., without menses for at least 12 consecutive months) or surgically sterile (i.e., those who underwent a hysterectomy with or without oophorectomy, fallopian tube ligation, and endometrial ablation).
10. Agreement to adhere to the following lifestyle compliance considerations:

    1. Refrain from consumption of grapefruit and any substance containing grapefruit for seven days prior to, during, and for seven days after the treatment day.
    2. Caffeine intake limited to 300 mg on treatment day (two 8-ounce cups).
    3. Abstain from alcohol for 24 hours prior to first dose of study medication.
    4. Refrain from any type of nicotine within 30 days prior to the screening visit and through the completion of the treatment day.

Exclusion Criteria:

1. Pregnancy, lactation, or positive serum pregnancy test at screening.
2. Known allergic reactions to scopolamine or other anticholinergics.
3. Currently prescribed any of the following medication types and used within the specified washout periods below:

   * belladonna alkaloids (washout 2 weeks),
   * antihistamines (including meclizine) (washout 2 weeks),
   * tricyclic antidepressants (washout 2 weeks),
   * muscle relaxants (washout 4 days) and
   * nasal decongestants (washout 4 days) (for Cohorts 1-4, and 6-16 only).
4. Hospitalization or significant surgery requiring hospital admittance within the past six months.
5. Treatment with another investigational drug or other intervention within the past 30 days.
6. Having donated blood or plasma or suffered significant blood loss within the past 30 days.
7. Use of nicotine within 30 days prior to the screening visit.
8. Having any of the following medical conditions within the last two years or if any of the following medical conditions were experienced more than two years ago and are deemed clinically significant by the PI or qualified designee:

   1. Significant gastrointestinal disorder, asthma, or seizure disorders.
   2. History of narrow-angle glaucoma.
   3. History of urinary retention or clinically significant symptomatic benign prostatic hypertrophy (BPH).
   4. History of moderate or severe substance use disorder.
   5. Nasal, nasal sinus, or nasal mucosa surgery (for Cohorts 1-4, and 6-16 only).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Describe the safety of Scopolamine HBr | The duration of participation for each subject will be approximately two weeks.
  Safety will be evaluated in terms of adverse events. Number of patients that report events of special interest as listed in the protocol.

CONTACTS AND LOCATIONS:
Overall Officials: David R Helton, Study Director — Repurposed Therapeutics, Inc.
Locations (1):
- Collaborative Neuroscience Network, LLC, Long Beach, California, United States